CLINICAL TRIAL: NCT01818258
Title: IMPAACT 1092: Phase IV Evaluation Of The Steady State Pharmacokinetics Of Zidovudine, Lamivudine, and Lopinavir/Ritonavir in Severely Malnourished HIV-1-Infected Children
Brief Title: IMPAACT P1092: Steady State PK in Malnourished HIV Infected Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPAACT P1092; U01AI068632 (NIH); 11689 (Other: DAIDS Study ID)
Record Dates: First submitted 2013-01-14; First posted 2013-03-26 (Estimated); Results first posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-07

CONDITIONS: HIV Positive; Malnourished
Keywords: HIV; Children; HAART; Malnourished
MeSH Terms: conditions — HIV Seropositivity; Malnutrition | interventions — Zidovudine; Lamivudine; Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Severe Malnutrition (Active Comparator): ZDV+3TC+LPV/r Zidovudine (ZDV, Retrovir®) 10 mg/ml oral syrup administered twice daily at WHO weight band dose for 48 weeks; Lamivudine (Epivir®, 3TC) 10 mg/ml for oral solution administered twice daily at WHO weight band dose for 48 weeks; Lopinavir/ritonavir (Kaletra®, LPV/r) 80/20 mg/ml oral solution administered twice daily at the WHO weight band dose for 48 weeks
  Interventions: Drug: ZDV+3TC+LPV/r
- Normal Nutrition/Mild Malnutrition (Active Comparator): ZDV+3TC+LPV/r Zidovudine (ZDV, Retrovir®) 10 mg/ml oral syrup administered twice daily at WHO weight band dose for 48 weeks; Lamivudine (Epivir®, 3TC) 10 mg/ml for oral solution administered twice daily at WHO weight band dose for 48 weeks; Lopinavir/ritonavir (Kaletra®, LPV/r) 80/20 mg/ml oral solution administered twice daily at the WHO weight band dose for 48 weeks
  Interventions: Drug: ZDV+3TC+LPV/r

INTERVENTIONS:
Drug: ZDV+3TC+LPV/r
  Other Names: Zidovudine; Retrovir; Lamivudine; Epivir; Lopinavir/ritonavir; Kaletra

SUMMARY:
Children living with HIV from sub-Saharan Africa often present with severe malnutrition. In severe malnutrition, metabolic and/or gut structural derangement may lead to inadequate antiretroviral (ARV) absorption and/or erratic drug levels. The greater surface area to weight ratio in severely malnourished children could also place them at higher risk of under dosing compared to children with mild to moderate malnutrition. However, limited data are available on the pharmacokinetics of ARVs in severely malnourished children. This study addressed this critical gap in knowledge by evaluating the PK of zidovudine (ZDV), lamivudine (3TC), and lopinavir/ritonavir (LPV/r) in severely malnourished children living with HIV, compared to children with normal nutrition to mild malnutrition living with HIV.

DETAILED DESCRIPTION:
P1092 was a prospective, non-randomized Phase IV open label study of antiretroviral drugs zidovudine (ZDV), lamivudine (3TC), and ritonavir boosted lopinavir (LPV/r) in children living with HIV aged 6 to less than 36 months grouped by nutritional status. The study's primary objectives were to characterize the pharmacokinetics (PK), safety, and tolerability of antiretroviral (ARV) regimens in severely acute malnourished (SAM) children following the initiation of nutritional rehabilitation and compare results to mildly malnourished or normally nourished children in order to determine if current recommended doses are optimal in severely malnourished children.

Two cohorts of children were enrolled based on nutritional status at screening: severely acute malnourished children and children with mild malnutrition or normal nutrition (non-SAM cohort). SAM participants were recruited from nutritional rehabilitation clinics while non-SAM participants were enrolled from HIV treatment centers. SAM participants were required to complete a 10 to 18 day nutritional rehabilitation program before entering the study. A World Health Organization (WHO, 2013) approach to management of SAM was used. All participants were to receive an antiretroviral regimen of ZDV+3TC+LPV/r. ARVs were dosed based on WHO weight band dosing and were to be administered twice per day in a pediatric liquid formulation. ZDV was allowed to be replaced with abacavir at the discretion of the site investigator/clinician in cases of grade 3 or higher hematologic toxicity on a ZDV-inclusive regimen or ZDV intolerance. Participants were followed for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of HIV-1 infection defined as positive results from two samples collected at different time points, using protocol-specified tests
* Meets WHO classification for severe malnutrition, normal nutrition status, or mild malnutrition
* Eligible for HAART defined by WHO 2013 pediatric guidelines
* Parent or legal guardian able and willing to provide signed informed consent, remain within the study area during the study period and agree to have subject followed at the clinical site
* Qualifying hematology and chemistry laboratory values obtained from specimens collected within the study-specific screening period
* For severely malnourished children: An inpatient in a nutrition rehabilitation unit. Clinical improvement after 10-18 days on nutrition rehabilitation defined as: Appetite returned and eating better - child shows interest in food even if does not complete amount given:
* No further weight loss
* Normalized sodium and potassium defined as severity grade 1 or lower
* No evidence of cardiac failure
* Loss of apathy and starting to play
* No hypothermia or pyrexia - temperature stable at >35.0 to <38.0° C (non-axillary) or >34.4 to <37.4° C (axillary)

For children with normal - mild malnutrition, clinical stability will be indicated by:

* Good appetite
* Normalized sodium and potassium defined as severity grade 1 or lower
* No hypothermia or pyrexia - temperature stable at >35.0 to <38.0° C (non-axillary) or >34.4 to <37.4° C (axillary)

Exclusion Criteria:

* Edematous malnutrition at the time of study entry
* ≥ Grade 3 respiratory distress or presence of cardio respiratory compromise within 3 days prior to entry
* Chemotherapy for malignancy
* Acute infection for which the child has received appropriate antimicrobial treatment for <5 days
* Tuberculosis disease
* Clinic hepatitis as evidenced by jaundice and hepatomegaly
* Taking any disallowed medications
* Any condition, situation, or clinical finding that in the opinion of the investigator would place the child at an unacceptable level of risk for injury, or render the child/caregiver(s) unable to meet the requirements of the study, interfere with study participation, or in the interpretation of study results.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2015-10-26 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maxensia O Owor, MBChB, MMED, MPH, Study Chair — International Maternal Pediatric Adolescent AIDS Clinical Trials Group
Locations (5):
- Malawi (2):
  - Blantyre CRS (30301), Blantyre
  - Malawi CRS (12001), Lilongwe
- Kilimanjaro Christian Medical Centre (5118), Moshi, Tanzania
- Makerere University-Johns Hopkins University (MUJHU) Research Collaboration (30293), Kampala, Uganda
- Harare Family Care (31890), Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No
* With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  * For what types of analyses? To achieve aims in the proposal approved by the IMPAACT Network.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/studies/submit-research-proposal. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data."

REFERENCES:
- [Result] Owor M, Tierney C, Ziemba L, Browning R, Moye J, Graham B, Reding C, Costello D, Norman J, Wiesner L, Hughes E, Whalen ME, Purdue L, Mmbaga BT, Kamthunzi P, Kawalazira R, Nathoo K, Bradford S, Coletti A, Aweeka F, Musoke P. Pharmacokinetics and Safety of Zidovudine, Lamivudine, and Lopinavir/Ritonavir in HIV-infected Children With Severe Acute Malnutrition in Sub-Saharan Africa: IMPAACT Protocol P1092. Pediatr Infect Dis J. 2021 May 1;40(5):446-452. doi: 10.1097/INF.0000000000003055. PMID 33464021
- [Derived] Bwakura-Dangarembizi M, Ziemba L, Tierney C, Reding C, Bone F, Bradford S, Costello D, Browning R, Moye J, Vhembo T, Ngocho JS, Mallewa M, Chinula L, Musoke P, Owor M. Micronutrients and nutritional status among children living with HIV with and without severe acute malnutrition: IMPAACT P1092. BMC Nutr. 2023 Nov 2;9(1):121. doi: 10.1186/s40795-023-00774-1. PMID 37919816
- See also: Signs/symptoms, laboratory events, and diagnoses were graded using the Division of AIDS (DAIDS) Table for Grading Severity of Adult and Pediatric Adverse Events, Corrected Version 2.0, November 2014. — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 52 participants, 25 in the Severe Acute Malnutrition (SAM) cohort and 27 in the non-SAM cohort, enrolled over a period of 12 months between October 26, 2015 and October 21, 2016. The SAM cohort was slower to enroll. Participants were enrolled from 5 sites in 4 African countries: Malawi, Tanzania, Uganda, and Zimbabwe.
Pre-assignment Details: Children with severe acute malnutrition (SAM) during the screening period were enrolled into the study 10-18 days after starting nutritional rehabilitation, and were required to show clinical improvement. SAM/non-SAM cohort assignments were determined during screening.
Groups:
- Severe Malnutrition Cohort: Severe Acute Malnutrition at Entry ZDV+3TC+LPV/r
- Normal Nutrition/Mild Malnutrition Cohort: Normal Nutrition or Mild Malnutrition at Entry ZDV+3TC+LPV/r
Period: Overall Study
Arm/Group | Severe Malnutrition Cohort | Normal Nutrition/Mild Malnutrition Cohort
Started | 25 | 27
Completed | 22 | 24
Not Completed | 3 | 3
Not completed — Death | 3 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Unable to Travel to Clinic | 0 | 1

BASELINE CHARACTERISTICS:
Population: All Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Severe Malnutrition Cohort | Normal Nutrition/Mild Malnutrition Cohort | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Mean (Standard Deviation); unit: months] | 19.4 (8.0) | 19.1 (8.5) | 19.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 16 | 13 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black Non-Hispanic | 25 | 27 | 52
Region of Enrollment [Count of Participants; unit: Participants]
  Tanzania | 7 | 9 | 16
  Uganda | 1 | 1 | 2
  Zimbabwe | 5 | 12 | 17
  Malawi | 12 | 5 | 17
World Health Organization (WHO) Weight-for-Height Z-Score [Mean (Standard Deviation); unit: Z-Score] — A Z-score indicates the number of standard deviations the measurement is away from the mean. A Z-score of 0 is equal to the mean of the reference population. Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population. The reference population was determined by the World Health Organization for children from 0 up to 5 years.
  Z-Score | -3.4 (0.8) | -0.7 (1.2) | -2.0 (1.7)
Mid-Upper Arm Circumference [Mean (Standard Deviation); unit: centimeters] | 11.1 (1.1) | 14.2 (1.6) | 12.7 (2.1)
Log10 Plasma HIV RNA Viral Load [Mean (Standard Deviation); unit: log 10 copies/mL] | 4.8 (1.2) | 5.2 (1.3) | 5.0 (1.3)
CD4 Percent [Mean (Standard Deviation); unit: percent] | 15.5 (8.8) | 24.5 (11.3) | 20.2 (11.1)
Nutritional Cohort Subgroup [Count of Participants; unit: Participants]
  Severe Malnutrition | 25 | 0 | 25
  Mild Malnutrition | 0 | 15 | 15
  Normal Nutrition | 0 | 12 | 12

OUTCOME MEASURES:

1. Primary Outcome: Grade 3 or Higher Adverse Events Through 24 Weeks
Description: Number (percent) of participants with at least one grade 3 or higher adverse event (AE) regardless of the relationship to study drugs.
Time Frame: From week 0 to week 24
Population: All participants who received at least one dose of study treatment (ZDV, 3TC, and LPV/r)
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Malnutrition Cohort | Normal Nutrition/Mild Malnutrition Cohort
Number analyzed (Participants) | 25 | 27
Participants | 13 | 10
Statistical Analysis 1: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Comparison for number who experienced at least one grade 3 or higher adverse event. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.40, Fisher Exact

2. Primary Outcome: Grade 3 or Higher Adverse Events Related to Study Drugs Through Week 24
Description: Number (percent) of participants with at least one Grade 3 or higher adverse event related to study drugs
Time Frame: From week 0 to week 24
Population: All participants who received at least one dose of study treatment (ZDV, 3TC, and LPV/r)
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Malnutrition Cohort | Normal Nutrition/Mild Malnutrition Cohort
Number analyzed (Participants) | 25 | 27
Participants | 6 | 7
Statistical Analysis 1: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Comparison for number who experienced at least one grade 3 or higher adverse event related to study treatment. Null hypothesis of no difference between cohorts; Test type: Superiority; p > 0.999, Fisher Exact

3. Primary Outcome: Steady-state Lopinavir Area Under the Curve
Description: Steady-state area under the curve (AUC) for Lopinavir (LPV)
Time Frame: 0, 1, 2, 4, 8, and 12 hours post-dose on 1, 12, and 24 weeks following study entry
Population: Participants with LPV AUC data at week 1 and at week 12 or 24
Measure: Geometric Mean (95% Confidence Interval); unit: ug*hours/mL
Arm/Group | Severe Malnutrition Cohort | Normal Nutrition/Mild Malnutrition Cohort
Number analyzed (Participants) | 22 | 23
ug*hours/mL
  Week 1 | 49.8 [28.5 to 87.2] | 64.8 [37.6 to 111.9]
  Week 12: number analyzed (Participants) | 21 | 23
  Week 12 | 53.0 [26.1 to 107.5] | 83.4 [60.4 to 115.0]
  Week 24: number analyzed (Participants) | 19 | 23
  Week 24 | 64.6 [28.3 to 147.5] | 79.4 [56.8 to 111.0]
Statistical Analysis 1: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 1 Comparison of LPV AUC between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.49, t-test, 2 sided; Geometric Mean Ratio = 0.77, 95% CI 2-sided [0.4 to 1.6] — Week 1 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition
Statistical Analysis 2: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 12 Comparison of LPV AUC between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.23, t-test, 2 sided; Geometric Mean Ratio = 0.64, 95% CI 2-sided [0.3 to 1.4] — Week 12 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition
Statistical Analysis 3: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 24 Comparison of LPV AUC between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.63, t-test, 2 sided; Geometric Mean Ratio = 0.81, 95% CI 2-sided [0.3 to 2.0] — Week 24 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition

4. Primary Outcome: Plasma Clearance of Lopinavir
Description: Steady-state plasma clearance (CL/F) of LPV
Time Frame: 0, 1, 2, 4, 8, and 12 hours post-dose on 1, 12, and 24 weeks following study entry
Population: Participants with LPV CL/F data at week 1 and at week 12 or 24
Measure: Geometric Mean (95% Confidence Interval); unit: L/hours
Arm/Group | Severe Malnutrition Cohort | Normal Nutrition/Mild Malnutrition Cohort
Number analyzed (Participants) | 22 | 23
L/hours
  LPV CL/F at Week 1 | 2.2 [1.2 to 3.9] | 2.0 [1.2 to 3.5]
  LPV CL/F at Week 12: number analyzed (Participants) | 21 | 23
  LPV CL/F at Week 12 | 2.3 [1.1 to 4.7] | 1.6 [1.2 to 2.3]
  LPV CL/F at Week 24: number analyzed (Participants) | 19 | 23
  LPV CL/F at Week 24 | 2.1 [0.9 to 4.8] | 1.7 [1.2 to 2.5]
Statistical Analysis 1: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 1 Comparison of LPV Clearance between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.89, t-test, 2 sided; Geometric Mean Ratio = 1.06, 95% CI 2-sided [0.5 to 2.3] — Week 1 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition
Statistical Analysis 2: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 12 Comparison of LPV clearance between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.37, t-test, 2 sided; Geometric Mean Ratio = 1.42, 95% CI 2-sided [0.7 to 3.1] — Week 12 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition
Statistical Analysis 3: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 24 Comparison of LPV clearance between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.63, t-test, 2 sided; Geometric Mean Ratio = 1.23, 95% CI 2-sided [0.5 to 2.9] — Week 24 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition

5. Primary Outcome: Steady-state Ritonavir Area Under the Curve
Description: Steady-state area under the curve (AUC) for Ritonavir (RTV)
Time Frame: 0, 1, 2, 4, 8, and 12 hours post-dose on 1, 12, and 24 weeks following study entry
Population: Participants with RTV AUC data at week 1 and at week 12 or 24
Measure: Geometric Mean (95% Confidence Interval); unit: ug*hours/mL
Arm/Group | Severe Malnutrition Cohort | Normal Nutrition/Mild Malnutrition Cohort
Number analyzed (Participants) | 22 | 23
ug*hours/mL
  RTV AUC Week 1 | 1.6 [1.0 to 2.5] | 2.1 [1.2 to 3.6]
  RTV AUC Week 12: number analyzed (Participants) | 21 | 23
  RTV AUC Week 12 | 1.8 [1.0 to 3.1] | 3.0 [2.1 to 4.5]
  RTV AUC Week 24: number analyzed (Participants) | 19 | 23
  RTV AUC Week 24 | 2.3 [1.3 to 4.3] | 3.0 [2.2 to 4.0]
Statistical Analysis 1: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 1 Comparison of RTV AUC between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.42, t-test, 2 sided; Geometric Mean Ratio = 0.76, 95% CI 2-sided [0.4 to 1.5] — Week 1 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition
Statistical Analysis 2: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 12 comparison of RTV AUC between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.11, t-test, 2 sided; Geometric Mean Ratio = 0.58, 95% CI 2-sided [0.3 to 1.1] — Week 12 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition
Statistical Analysis 3: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 24 comparison of RTV AUC between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.44, t-test, 2 sided; Geometric Mean Ratio = 0.77, 95% CI 2-sided [0.4 to 1.5] — Week 24 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition

6. Primary Outcome: Plasma Clearance of Ritonavir
Description: Steady-state plasma clearance (CL/F) of RTV
Time Frame: 0, 1, 2, 4, 8, and 12 hours post-dose on 1, 12, and 24 weeks following study entry
Population: Participants with RTV CL/F data at week 1 and at week 12 or 24
Measure: Geometric Mean (95% Confidence Interval); unit: L/hours
Arm/Group | Severe Malnutrition Cohort | Normal Nutrition/Mild Malnutrition Cohort
Number analyzed (Participants) | 22 | 23
L/hours
  RTV CL/F at Week 1 | 16.9 [10.5 to 27.2] | 15.8 [9.2 to 27.2]
  RTV CL/F at Week 12: number analyzed (Participants) | 21 | 23
  RTV CL/F at Week 12 | 17.3 [9.6 to 31.0] | 11.2 [7.6 to 16.6]
  RTV CL/F at Week 24: number analyzed (Participants) | 19 | 23
  RTV CL/F at Week 24 | 14.8 [8.1 to 27.2] | 11.5 [8.4 to 15.7]
Statistical Analysis 1: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 1 comparison of RTV clearance between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.84, t-test, 2 sided; Geometric Mean Ratio = 1.07, 95% CI 2-sided [0.5 to 2.2] — Week 1 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition
Statistical Analysis 2: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 12 comparison of RTV clearance between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.21, t-test, 2 sided; Geometric Mean Ratio = 1.54, 95% CI 2-sided [0.8 to 3.1] — Week 12 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition
Statistical Analysis 3: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 24 comparison of RTV clearance between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.44, t-test, 2 sided; Geometric Mean Ratio = 1.29, 95% CI 2-sided [0.7 to 2.5] — Week 24 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition

7. Primary Outcome: Steady-state Lamivudine Area Under the Curve
Description: Steady-state area under the curve (AUC) of Lamivudine (3TC)
Time Frame: 0, 1, 2, 4, 8, and 12 hours post-dose on 1, 12, and 24 weeks following study entry
Population: Participants with 3TC AUC data at week 1 and at week 12 or 24
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hours/mL
Arm/Group | Severe Malnutrition Cohort | Normal Nutrition/Mild Malnutrition Cohort
Number analyzed (Participants) | 21 | 21
ng*hours/mL
  3TC AUC at Week 1 | 4,245.0 [2,959.3 to 6,089.3] | 5,520.2 [3,981.4 to 7,653.7]
  3TC AUC at Week 12: number analyzed (Participants) | 20 | 21
  3TC AUC at Week 12 | 4,365.5 [2,743.6 to 6,946.4] | 7,233.0 [5,896.4 to 8,872.6]
  3TC AUC at Week 24: number analyzed (Participants) | 18 | 20
  3TC AUC at Week 24 | 6,359.0 [5,221.9 to 7,743.8] | 5,849.2 [3,453.5 to 9,907.0]
Statistical Analysis 1: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 1 comparison of 3TC AUC between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.27, t-test, 2 sided; Geometric Mean Ratio = 0.77, 95% CI 2-sided [0.5 to 1.2] — Week 1 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition
Statistical Analysis 2: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 12 comparison of 3TC AUC between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.047, t-test, 2 sided; Geometric Mean Ratio = 0.60, 95% CI 2-sided [0.4 to 1.0] — Week 12 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition
Statistical Analysis 3: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 24 comparison of 3TC AUC between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.76, t-test, 2 sided; Geometric Mean Ratio = 1.09, 95% CI 2-sided [0.6 to 1.9] — Week 24 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition

8. Primary Outcome: Plasma Clearance of Lamivudine
Description: Steady-state plasma clearance (CL/F) of Lamivudine (3TC)
Time Frame: 0, 1, 2, 4, 8, and 12 hours post-dose on 1, 12, and 24 weeks following study entry
Population: Participants with 3TC CL/F data at week 1 and at week 12 or 24
Measure: Geometric Mean (95% Confidence Interval); unit: L/hours
Arm/Group | Severe Malnutrition Cohort | Normal Nutrition/Mild Malnutrition Cohort
Number analyzed (Participants) | 21 | 21
L/hours
  3TC CL/F at Week 1 | 8.7 [6.0 to 12.7] | 8.4 [6.2 to 11.5]
  3TC CL/F at Week 12: number analyzed (Participants) | 20 | 21
  3TC CL/F at Week 12 | 9.5 [5.9 to 15.4] | 6.8 [5.7 to 8.1]
  3TC CL/F at Week 24: number analyzed (Participants) | 18 | 20
  3TC CL/F at Week 24 | 7.5 [6.2 to 9.0] | 8.8 [5.3 to 14.7]
Statistical Analysis 1: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 1 comparison of 3TC clearance between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.89, t-test, 2 sided; Geometric Mean Ratio = 0.0, 95% CI 2-sided [-0.4 to 0.5] — Week 1 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition
Statistical Analysis 2: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 12 comparison of 3TC clearance between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.18, t-test, 2 sided; Geometric Mean Ratio = 1.40, 95% CI 2-sided [0.8 to 2.3] — Week 12 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition
Statistical Analysis 3: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 24 comparison of 3TC clearance between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.53, t-test, 2 sided; Geometric Mean Ratio = 0.85, 95% CI 2-sided [0.5 to 1.4] — Week 24 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition

9. Primary Outcome: Steady-state Zidovudine Area Under the Curve
Description: Steady-state area under the curve (AUC) of zidovudine (ZDV)
Time Frame: 0, 1, 2, 4, 8, and 12 hours post-dose on 1, 12, and 24 weeks following study entry
Population: Participants with ZDV AUC data at week 1 and at week 12 or 24
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hours/mL
Arm/Group | Severe Malnutrition Cohort | Normal Nutrition/Mild Malnutrition Cohort
Number analyzed (Participants) | 15 | 16
ng*hours/mL
  ZDV AUC at Week 1 | 2,261.0 [1,652.0 to 3,094.4] | 1,774.0 [1,079.6 to 2,915.1]
  ZDV AUC at Week 12: number analyzed (Participants) | 12 | 16
  ZDV AUC at Week 12 | 1,826.0 [977.8 to 3,410.0] | 1,335.7 [758.5 to 2,352.2]
  ZDV AUC at Week 24: number analyzed (Participants) | 13 | 15
  ZDV AUC at Week 24 | 2,449.7 [2,053.5 to 2,922.5] | 1,609.3 [1,306.7 to 1,981.9]
Statistical Analysis 1: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 1 comparison of ZDV AUC between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.39, t-test, 2 sided; Geometric Mean Ratio = 1.27, 95% CI 2-sided [0.7 to 2.2] — Week 1 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition
Statistical Analysis 2: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 12 comparison of ZDV AUC between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.43, t-test, 2 sided; Geometric Mean Ratio = 1.37, 95% CI 2-sided [0.6 to 3.0] — Week 12 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition
Statistical Analysis 3: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 24 comparison of ZDV AUC between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.003, t-test, 2 sided; Geometric Mean Ratio = 1.52, 95% CI 2-sided [1.2 to 2.0] — Week 24 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition

10. Primary Outcome: Plasma Clearance of Zidovudine
Description: Steady-state plasma clearance (CL/F) of Zidovudine (ZDV)
Time Frame: 0, 1, 2, 4, 8, and 12 hours post-dose on 1, 12, and 24 weeks following study entry
Population: Participants with ZDV CL/F data at week 1 and at week 12 or 24
Measure: Geometric Mean (95% Confidence Interval); unit: L/hours
Arm/Group | Severe Malnutrition Cohort | Normal Nutrition/Mild Malnutrition Cohort
Number analyzed (Participants) | 15 | 16
L/hours
  ZDV CL/F at Week 1 | 34.8 [24.4 to 49.5] | 58.3 [34.8 to 97.9]
  ZDV CL/F at Week 12: number analyzed (Participants) | 12 | 16
  ZDV CL/F at Week 12 | 48.8 [24.8 to 95.8] | 81.8 [44.9 to 148.9]
  ZDV CL/F at Week 24: number analyzed (Participants) | 13 | 15
  ZDV CL/F at Week 24 | 40.8 [33.0 to 50.4] | 64.0 [51.7 to 79.1]
Statistical Analysis 1: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 1 comparison of ZDV clearance between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.090, t-test, 2 sided; Geometric Mean Ratio = 0.60, 95% CI 2-sided [0.3 to 1.1] — Week 1 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition
Statistical Analysis 2: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 12 comparison of ZDV clearance between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.23, t-test, 2 sided; Geometric Mean Ratio = 0.60, 95% CI 2-sided [0.3 to 1.4] — Week 12 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition
Statistical Analysis 3: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 24 comparison of ZDV clearance between cohorts. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.0003, t-test, 2 sided; Geometric Mean Ratio = 0.64, 95% CI 2-sided [0.5 to 0.8] — Week 24 Geometric Mean Ratio of Severe Malnutrition/Normal Nutrition/Mild Malnutrition

11. Secondary Outcome: Minimum Trough Concentration (Ctrough) of Lopinavir
Description: Count (%) of participants with minimum trough concentration (Ctrough) of steady-state Lopinavir >= 1 ug/mL
Time Frame: Measured 0, 1, 2, 4, 8, and 12 hours post-dose on 1, 4, 8, 12, 16, 24, 36 and 48 weeks following study entry
Population: Participants with minimum trough concentration of LPV data
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Malnutrition Cohort | Normal Nutrition/Mild Malnutrition Cohort
Number analyzed (Participants) | 24 | 25
Participants
  Week 1 | 12 | 21
  Week 4: number analyzed (Participants) | 23 | 24
  Week 4 | 14 | 18
  Week 8: number analyzed (Participants) | 22 | 24
  Week 8 | 13 | 18
  Week 12: number analyzed (Participants) | 22 | 24
  Week 12 | 17 | 18
  Week 16: number analyzed (Participants) | 21 | 22
  Week 16 | 11 | 15
  Week 24: number analyzed (Participants) | 20 | 23
  Week 24 | 14 | 19
  Week 36: number analyzed (Participants) | 20 | 24
  Week 36 | 16 | 19
  Week 48: number analyzed (Participants) | 18 | 22
  Week 48 | 16 | 18
Statistical Analysis 1: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Odds ratio (SAM/non-SAM) of Ctrough >=1 ug/mL from entry through 48 weeks from repeated measures mixed model, with the null hypothesis that the odds ratio is equal to zero (no difference between cohorts in odds of Ctrough >=1 ug/mL); Test type: Superiority; p = 0.17, Mixed Models Analysis; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.22 to 1.29] — Odds Ratio (SAM/non-SAM) for Lopinavir Ctrough >= 1 ug/mL through 48 weeks

12. Secondary Outcome: Free Fraction of LPV at Hour 2 Post Dose
Description: Free fraction of steady-state lopinavir at 2 hours post dose
Time Frame: Weeks 1, 12 and 24
Population: Participants with LPV free fraction data available
Measure: Mean (Standard Deviation); unit: Percent of Unbound LPV
Arm/Group | Severe Malnutrition Cohort | Normal Nutrition/Mild Malnutrition Cohort
Number analyzed (Participants) | 9 | 14
Percent of Unbound LPV
  Week 1: number analyzed (Participants) | 6 | 14
  Week 1 | 0.8 (0.8) | 3.2 (2.3)
  Week 12: number analyzed (Participants) | 9 | 10
  Week 12 | 2.2 (1.0) | 6.0 (3.8)
  Week 24: number analyzed (Participants) | 5 | 4
  Week 24 | 3.1 (2.8) | 2.1 (0.6)
Statistical Analysis 1: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 1 comparison of LPV free faction. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.003, t-test, 2 sided; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-3.9 to -0.9] — Severe Malnutrition Cohort - Normal Nutrition/Mild Malnutrition for Week 1 Free Fraction (%) of LPV
Statistical Analysis 2: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 12 comparison of LPV free faction. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.011, t-test, 2 sided; Mean Difference (Final Values) = -3.8, 95% CI 2-sided [-6.6 to -1.1] — Severe Malnutrition - Normal Nutrition/Mild Malnutrition for Week 12 Free Fraction (%) of LPV
Statistical Analysis 3: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 24 comparison of LPV free faction. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.46, t-test, 2 sided; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-2.4 to 4.4] — Severe Malnutrition - Normal Nutrition/Mild Malnutrition for Week 24 Free Fraction (%) of LPV

13. Secondary Outcome: Change in HIV Viral Load From Baseline
Description: Change from baseline in plasma HIV RNA viral load
Time Frame: Weeks 0, 12, 24, 36 and 48
Population: Participants with data at baseline and timepoint of interest (week 12, 24, 36, or 48)
Measure: Mean (95% Confidence Interval); unit: log10 copies/mL
Arm/Group | Severe Malnutrition Cohort | Normal Nutrition/Mild Malnutrition Cohort
Number analyzed (Participants) | 22 | 23
log10 copies/mL
  Change in Log10 Viral Load between Baseline and Week 12 | -1.4 [-2.1 to -0.7] | -2.1 [-2.8 to -1.4]
  Change in Log10 Viral Load between Baseline and Week 24: number analyzed (Participants) | 21 | 22
  Change in Log10 Viral Load between Baseline and Week 24 | -1.7 [-2.6 to -0.9] | -2.5 [-3.3 to -1.7]
  Change in Log10 Viral Load between Baseline and Week 36: number analyzed (Participants) | 21 | 23
  Change in Log10 Viral Load between Baseline and Week 36 | -1.8 [-2.5 to -1.0] | -2.5 [-3.2 to -1.8]
  Change in Log10 Viral Load between Baseline and Week 48: number analyzed (Participants) | 21 | 22
  Change in Log10 Viral Load between Baseline and Week 48 | -1.8 [-2.5 to -1.1] | -2.6 [-3.4 to -1.9]
Statistical Analysis 1: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Difference in cohorts of change in log10 plasma HIV viral load from baseline to week 12. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.15, t-test, 2 sided; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-0.3 to 1.7] — Direction of comparison: Severe Malnutrition - Normal Nutrition/Mild Malnutrition
Statistical Analysis 2: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Difference in cohorts of change in log10 plasma HIV viral load from baseline to week 24. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.20, t-test, 2 sided; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-0.4 to 1.8] — Direction of comparison: Severe Malnutrition - Normal Nutrition/Mild Malnutrition
Statistical Analysis 3: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Difference in cohorts of change in log10 plasma HIV viral load from baseline to week 36. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.13, t-test, 2 sided; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-0.2 to 1.8] — Direction of comparison: Severe Malnutrition - Normal Nutrition/Mild Malnutrition
Statistical Analysis 4: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Difference in cohorts of change in log10 plasma HIV viral load from baseline to week 48. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.089, t-test, 2 sided; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-0.1 to 1.8] — Direction of comparison: Severe Malnutrition - Normal Nutrition/Mild Malnutrition

14. Secondary Outcome: HIV Viral Load <400 Copies/mL
Description: Count (%) of participants with plasma HIV RNA viral load <400 copies/mL
Time Frame: Baseline and weeks 12, 24, and 48
Population: Participants with data at baseline and timepoint of interest (week 12, 24, or 48)
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Malnutrition Cohort | Normal Nutrition/Mild Malnutrition Cohort
Number analyzed (Participants) | 25 | 27
Participants
  Baseline | 2 | 2
  Week 12: number analyzed (Participants) | 23 | 24
  Week 12 | 8 | 14
  Week 24: number analyzed (Participants) | 22 | 23
  Week 24 | 11 | 18
  Week 48: number analyzed (Participants) | 22 | 23
  Week 48 | 11 | 18
Statistical Analysis 1: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Baseline Comparison, with null hypothesis of no difference between cohorts; Test type: Superiority; p > 0.999, Fisher Exact
Statistical Analysis 2: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 12 Comparison, with null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.15, Fisher Exact
Statistical Analysis 3: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 24 Comparison, with null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.065, Fisher Exact
Statistical Analysis 4: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Week 48 Comparison, with null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.065, Fisher Exact

15. Secondary Outcome: Change in CD4 Percent
Description: Change in CD4 percent from baseline
Time Frame: Weeks 0, 12, 24, 36 and 48
Population: Participants with CD4 percent data at baseline and timepoint of interest (week 12, 24, 36, or 48)
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | Severe Malnutrition Cohort | Normal Nutrition/Mild Malnutrition Cohort
Number analyzed (Participants) | 23 | 24
percent
  Change in CD4 Percent at Week 12 | 3.3 [0.0 to 6.5] | 3.0 [0.2 to 5.8]
  Change in CD4 Percent at Week 24: number analyzed (Participants) | 21 | 23
  Change in CD4 Percent at Week 24 | 9.3 [5.0 to 13.7] | 6.8 [4.0 to 9.6]
  Change in CD4 Percent at Week 36: number analyzed (Participants) | 21 | 24
  Change in CD4 Percent at Week 36 | 10.3 [6.1 to 14.4] | 7.1 [4.7 to 9.5]
  Change in CD4 Percent at Week 48: number analyzed (Participants) | 22 | 24
  Change in CD4 Percent at Week 48 | 12.7 [8.3 to 17.1] | 6.7 [4.2 to 9.1]
Statistical Analysis 1: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Difference in cohorts of change in CD4 percent from baseline to week 12. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.89, t-test, 2 sided; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-3.9 to 4.4] — Direction of comparison: Severe Malnutrition - Normal Nutrition/Mild Malnutrition
Statistical Analysis 2: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Difference in cohorts of change in CD4 percent from baseline to week 24. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.31, t-test, 2 sided; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [-2.5 to 7.6] — Direction of comparison: Severe Malnutrition - Normal Nutrition/Mild Malnutrition
Statistical Analysis 3: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Difference in cohorts of change in CD4 percent from baseline to week 36. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.18, t-test, 2 sided; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [-1.5 to 7.8] — Direction of comparison: Severe Malnutrition - Normal Nutrition/Mild Malnutrition
Statistical Analysis 4: Comparison: Severe Malnutrition Cohort vs Normal Nutrition/Mild Malnutrition Cohort; Difference between cohorts of change in CD4 percent from baseline to week 48. Null hypothesis of no difference between cohorts; Test type: Superiority; p = 0.018, t-test, 2 sided; Mean Difference (Final Values) = 6.1, 95% CI 2-sided [1.1 to 11.0] — Direction of comparison: Severe Malnutrition - Normal Nutrition/Mild Malnutrition

16. Secondary Outcome: Change in WHO Weight-for-height Z-score
Description: Change in WHO weight-for-height Z-score from entry. A Z-score indicates the number of standard deviations the measurement is away from the mean. A Z-score of 0 is equal to the mean of the reference population. Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population. The reference population was determined by the World Health Organization for children from 0 up to 5 years.
Time Frame: Weeks 0, 24, and 48
Population: Participants with weight and height data available
Measure: Mean (95% Confidence Interval); unit: Z-Score
Arm/Group | Severe Malnutrition Cohort | Normal Nutrition/Mild Malnutrition Cohort
Number analyzed (Participants) | 25 | 27
Z-Score
  Week 24: number analyzed (Participants) | 22 | 23
  Week 24 | 2.3 [1.8 to 2.9] | 0.1 [-0.3 to 0.5]
  Week 48: number analyzed (Participants) | 22 | 24
  Week 48 | 2.7 [2.1 to 3.4] | 0.4 [-0.1 to 0.8]
Statistical Analysis 1: Comparison: Severe Malnutrition Cohort; Null hypothesis: change in WHO weight-for-height Z-score from entry to week 24 equal to 0; Test type: Superiority; p < 0.0001, t-test, 2 sided; Mean = 2.34, 95% CI 2-sided [1.77 to 2.91]
Statistical Analysis 2: Comparison: Severe Malnutrition Cohort; Null hypothesis: change in WHO weight-for-height Z-score from entry to week 48 equal to 0; Test type: Superiority; p < 0.0001, t-test, 2 sided; Mean = 2.73, 95% CI 2-sided [2.09 to 3.37]

17. Secondary Outcome: Change in Mid-upper Arm Circumference
Description: Change in mid-upper arm circumference (MUAC) from entry
Time Frame: Weeks 0, 24, and 48
Population: Participants with MUAC data available
Measure: Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Severe Malnutrition Cohort | Normal Nutrition/Mild Malnutrition Cohort
Number analyzed (Participants) | 23 | 24
centimeters
  Week 24: number analyzed (Participants) | 22 | 23
  Week 24 | 2.6 [2.0 to 3.3] | 1.2 [0.8 to 1.6]
  Week 48: number analyzed (Participants) | 22 | 24
  Week 48 | 3.5 [2.8 to 4.2] | 1.6 [1.2 to 2.0]
Statistical Analysis 1: Comparison: Severe Malnutrition Cohort; Null hypothesis: change in MUAC from entry to week 24 equal to 0; Test type: Superiority; p < 0.0001, t-test, 2 sided; Mean = 2.63, 95% CI 2-sided [1.96 to 3.28]
Statistical Analysis 2: Comparison: Severe Malnutrition Cohort; Null hypothesis: change in MUAC from entry to week 48 equal to 0; Test type: Superiority; p < 0.0001, t-test, 2 sided; Mean = 3.53, 95% CI 2-sided [2.83 to 4.24]

ADVERSE EVENTS:
Time Frame: From study entry to study completion at Week 48 or premature study discontinuation
Description: Serious Adverse Event (SAE) Reporting Category [v2.0 of the DAIDS expedited adverse event Manual] was used. Study agents for which relationship assessments were required: ZDV, 3TC, LPV/r and abacavir. Other events reported in an expedited fashion included malignancies, seizures and Grade 3/4 hepatotoxicities, and Grade 3/4 related toxicities where a relationship to study drug could not be ruled out. Events were summarized if onset was on or after entry.
Groups:
- Severe Malnutrition: Severe Acute Malnutrition at Entry ZDV+3TC+LPV/r
- Normal Nutrition/Mild Malnutrition: Normal Nutrition or Mild Malnutrition at Entry ZDV+3TC+LPV/r
Arm/Group | Severe Malnutrition | Normal Nutrition/Mild Malnutrition
All-Cause Mortality (participants affected / at risk) | 3/25 | 0/27
Serious Adverse Events (participants affected / at risk) | 9/25 | 5/27
Other Adverse Events (participants affected / at risk) | 25/25 | 25/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Severe Malnutrition (N=25) | Normal Nutrition/Mild Malnutrition (N=27)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Haemoglobin decreased (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 3 | 0
Malnutrition (Metabolism and nutrition disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Severe Malnutrition (N=25) | Normal Nutrition/Mild Malnutrition (N=27)
Anaemia (Blood and lymphatic system disorders) | 5 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 4 | 5
Splenomegaly (Blood and lymphatic system disorders) | 2 | 1
Otorrhoea (Ear and labyrinth disorders) | 4 | 3
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 4 | 3
Eye discharge (Eye disorders) | 4 | 5
Ocular hyperaemia (Eye disorders) | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 11 | 6
Oral disorder (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 1
Vomiting (Gastrointestinal disorders) | 8 | 5
Pyrexia (General disorders) | 11 | 10
Conjunctivitis (Infections and infestations) | 3 | 3
Gastroenteritis (Infections and infestations) | 5 | 2
Impetigo (Infections and infestations) | 4 | 0
Oral candidiasis (Infections and infestations) | 6 | 1
Otitis media acute (Infections and infestations) | 6 | 5
Plasmodium falciparum infection (Infections and infestations) | 6 | 5
Pneumonia bacterial (Infections and infestations) | 3 | 5
Tinea faciei (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 2
Alanine aminotransferase increased (Investigations) | 5 | 3
Aspartate aminotransferase increased (Investigations) | 6 | 3
Blood albumin decreased (Investigations) | 16 | 10
Blood bicarbonate decreased (Investigations) | 23 | 20
Blood cholesterol increased (Investigations) | 3 | 2
Blood glucose decreased (Investigations) | 5 | 4
Blood glucose increased (Investigations) | 2 | 1
Blood potassium decreased (Investigations) | 2 | 0
Blood potassium increased (Investigations) | 10 | 8
Blood sodium decreased (Investigations) | 12 | 15
Blood triglycerides increased (Investigations) | 1 | 4
Haemoglobin decreased (Investigations) | 22 | 21
Neutrophil count decreased (Investigations) | 7 | 17
Platelet count decreased (Investigations) | 3 | 3
Weight decreased (Investigations) | 7 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 21 | 6
Poor feeding infant (Metabolism and nutrition disorders) | 5 | 1
Underweight (Metabolism and nutrition disorders) | 6 | 0
Selective eating disorder (Psychiatric disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Papule (Skin and subcutaneous tissue disorders) | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 3
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 3
Pallor (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Children with moderate malnutrition were not enrolled in the study by design

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT01818258/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT01818258/SAP_001.pdf